CLINICAL TRIAL: NCT00987662
Title: Double Blind Study of Irbesartan vs. Amlodipine in Obese Hypertensive Subjects- The OBI Study
Brief Title: Irbesartan Versus Amlodipine: The OBI Study
Acronym: OBI
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: no funding
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Kotsis Vasilios/Prof, Papageorgiou hospital hypertension/24h ABPM center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: AUTH170909
Record Dates: First submitted 2009-09-30; First posted 2009-10-01 (Estimated); Last update posted 2014-02-11 (Estimated); Status verified 2009-09

CONDITIONS: Obesity; Hypertension
Keywords: irbesartan; amlodipine; obesity; ambulatory blood pressure monitoring; new onset diabetes
MeSH Terms: conditions — Obesity; Hypertension | interventions — Irbesartan; Amlodipine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Irbesartan (Active Comparator): Treatment with irbesartan 300mg for 4 weeks. IF ABP>135/85 mmHg add HCZ 12.5 mg.
  Interventions: Drug: Irbesartan
- Amplodipine (Active Comparator): Treatment with amlodipine 10 mg for 4 weeks. If BP>135/85 mmHg add hydrochlorothiazide 12.5 mg
  Interventions: Drug: Amlodipine

INTERVENTIONS:
Drug: Irbesartan — Treatment with irbesartan 300mg for 4 weeks. IF ABP>135/85 mmHg add hydrochlorothiazide 12.5 mg.
  Arms: Irbesartan
Drug: Amlodipine — Treatment with amlodipine 10 mg for 4 weeks. If ABP>135/85 mmHg add hydrochlorothiazide 12.5 mg
  Arms: Amplodipine

SUMMARY:
Objective:

1. To study the effectiveness of irbesartan 300mg and amlodipine 10 mg in 24h ambulatory blood pressure values in obese subjects
2. To study the drug specific effect in arterial stiffness
3. To study possible drug mechanisms in obesity (reduction of central adiposity and changing the ratio of leptin to adiponectin)

DETAILED DESCRIPTION:
Study Objectives

1. Primary:

   * Reduction of 24h BP in obese hypertensives
   * Reduction in arterial stiffness
2. Secondary

   * Drug specific effect on new onset of diabetes
   * Drug specific effect on reduction in central fat deposition and the leptin to adiponectin ratio

Study design

Study drugs: Irbesartan 300mg vs. amlodipine 10mg

Tx duration and follow-up: 12 months

Collected data:

* 24h SBP and DBP in time 0, 1, 12.
* Pulse wave velocity in time 0,1,12.
* Central obesity (total, visceral, abdominal fat) in time 0,1,12.
* Leptin/adiponectin in time 0,1,12.
* BMI, waist/hip ratio in time 0,1, 12.
* Glu, HbA1c, insulin in time 0, 1,12.
* K, Na, Cr, BUN, Chol, Tg, HDL, LDL,ALT, AST in time 0, 1,12. Number of patients: The reduction in mean SBP expected to be 15 mmHg. Previous studies from our group reported an 14mmHg SD for mean SBP. The sample size required at the two sided 5% significance level and 80% power is 40 patients (Lehr's formula)

Number of centers: 1

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 60 years.
2. All patients are going to give their informed consent to participate in the study.
3. Stage I hypertension.
4. BMI > 30.

Exclusion Criteria:

1. Known oversensitiveness,
2. Chronic renal disease (GFR < 50 ml/min) or ESRD,
3. Heart or respiratory failure, OR
4. Recent MI, shock, liver deficiency (ALT or AST > 3 times normal and pregnancy or lactation.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2012-01; Primary Completion 2013-01 (Estimated); Study Completion 2014-01 (Estimated)

PRIMARY OUTCOMES:
Reduction of 24h BP and arterial stiffness in obese hypertensives | 12

SECONDARY OUTCOMES:
New onset of diabetes | 12
Drug specific effect on reduction in central fat deposition and the leptin to adiponectin ratio | 12

CONTACTS AND LOCATIONS:
Overall Officials: Vasilios Kotsis, Prof, Study Chair — AUTH
Locations (1):
- Hypertension-24h ABPM Center Papageorgiou Hospital, Thessaloniki, Greece